CLINICAL TRIAL: NCT00751894
Title: Haematopoietic Progenitor Cell Mobilization in Children With Malignancies: Evaluation of Pegfilgrastim at 200µg/kg After Chemotherapy
Brief Title: Pegfilgrastim for Stem Cell Mobilization in Children (Meg-5)
Acronym: MEG-5
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Amgen (Industry)
Responsible Party: Dr Etienne MERLIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0041
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Solid Malignancies
Keywords: Children; cancer; Bone marrow transplantation; Stem cell mobilization; G-CSF; Children with solid malignancies
MeSH Terms: conditions — Neoplasms | interventions — pegfilgrastim

INTERVENTIONS:
Drug: Pegfilgrastim (Neulasta, Amgen) — sequential Bayesian study

SUMMARY:
Hypothesis : pegfilgrastim at 200 µg/kg between 12 and 18 days after previous chemotherapy provides an efficient stem cell mobilization in children with malignancies Design: phase 2 study. Judgment criterion: percentage of children achieving at least 5x10e6 CD34 cells with a standard apheresis (less than 3 blood volume processed

DETAILED DESCRIPTION:
Patients: consecutively referred for HSC mobilization. 12 to 18 days after the previous chemotherapy. No haematological growth factor during the 8 previous days.

Mobilization: one sc injection of 200 µg/kg pegfilgrastim (Neulasta, Amgen) Evaluation during the study: CD34 circulating cells from day 3 to day 7 ; AE recording Judgment criterion: percentage of children achieving at least 5x10e6 CD34 cells with a standard apheresis (less than 3 blood volume processed) Analysis: sequential Bayesian study

ELIGIBILITY:
Inclusion Criteria:

* 0 to 18 years
* solid malignancy
* Lansky score >70%
* 12 to 18 days since the beginning of the last chemotherapy cycle
* no administration of any hematopoietic growth factor in the previous 8 days

Exclusion Criteria:

* clinical or biological conditions precluding the mobilization or collection procedure

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)

PRIMARY OUTCOMES:
percentage of children achieving at least 5x10e6 CD34 cells with a standard apheresis (less than 3 blood volume processed) | less than 3 blood volume processed

SECONDARY OUTCOMES:
Side effects Number of apheresis required to achieved a graft of at least 5x10e6 CD34 cells | at least 5*10e6CD34cells

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Merlin, DR, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France